CLINICAL TRIAL: NCT05168774
Title: A Pilot Investigator Initiated Study to Evaluate the Safety, Tolerability and Efficacy of Elamipretide in the Treatment of Advanced Symptoms of Friedreich Ataxia (FRDA)
Brief Title: FRDA Investigator Initiated Study (IIS) With Elamipretide
Acronym: ELViS-FA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Friedreich's Ataxia Research Alliance (Other); Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Principal Investigator, David Lynch, Professor of Neurology in Pediatrics at the Children's Hospital of Philadelphia, Children's Hospital of Philadelphia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-018049; SPIFA-101 (Other: Stealth Biotherapeutics, Inc.)
Expanded Access: NCT04689360 (Available)
Record Dates: First submitted 2021-12-09; First posted 2021-12-23 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Friedreich Ataxia
Keywords: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low Dose (20-30mg) (Experimental): Subjects will receive daily subcutaneous (SC) dosing of Elamipretide (20-30 mg) for 52 weeks
  Interventions: Drug: Elamipretide
- High Dose (40-60 mg) (Experimental): Subjects will receive daily subcutaneous (SC) dosing of Elamipretide (40-60 mg) for 52 weeks
  Interventions: Drug: Elamipretide

INTERVENTIONS:
Drug: Elamipretide — Elamipretide is a tetra peptide with limited blood brain barrier penetration being developed for use in a variety of mitochondrial disorders, including FRDA, mitochondrial myopathy and Barth Syndrome.
  Other Names: MTP-131; SS-31

SUMMARY:
To evaluate the safety, tolerability, and activity of Elamipretide in treating vision loss in Friedreich Ataxia (FRDA).

DETAILED DESCRIPTION:
To evaluate the effect of high dose (40-60mg) versus low dose (20-30mg) Elamipretide on high contrast visual acuity in FRDA compared to baseline at 52 weeks with the option to extend for an additional 52 weeks if there are objective signs of clinical improvement on primary or secondary endpoints. The interim analysis will be based on data from a 36-week visit. For subjects worse than 20/800 at study start, they will be followed using low vision alternatives only.

ELIGIBILITY:
Inclusion Criteria:

1. Genetically confirmed FRDA (point mutations allowed).
2. Age >16 years.
3. Disease onset before 18 years of age.
4. If female, the subject is not pregnant or lactating or intending to become pregnant before, during, or within 30 days after the last dose of study drug. Female subjects of child-bearing potential must have a negative serum pregnancy test result at Screening, a negative urine pregnancy test result at Baseline.
5. All subjects must agree to use a reliable method of contraception throughout the study and for 30 days after the last dose of study drug. Male subjects should not father a baby during the study or for at least 30 days after the last dose of study drug.
6. All concomitant medications (including over-the-counter medications), vitamins, and supplements must be at stable doses for 30 days prior to study entry and kept stable throughout the study to the best of their ability.
7. Visual acuity (VA) worse than 20/40 (binocular) on the basis of FRDA. Must not be correctable by refraction, or subjects must have sufficient physical exam findings of optic neuropathy (funduscopic, visual fields, or retinal ganglion cell loss) to justify the primary diagnosis of FRDA related optic neuropathy

   Or
8. Ejection Fraction (EF) less than 50% at last evaluation (within 1 year before screening), with a history consistent with cardiomyopathy from FRDA, and VA 20/25- 20/40.

Exclusion Criteria:

1. Any unstable illness that in the investigator's opinion precludes participation in the study.
2. Use of any investigational product within 30 days prior to Screening.
3. A history of substance abuse.
4. Diagnosis of active HIV or Hepatitis B or C infection.
5. Presence of severe renal disease (eGFR <30 mL/min) or hepatic disease [aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2x the upper limit of normal] as evidenced by laboratory results at Screening.
6. Clinically significant abnormal white blood cell count (ANC <1500), hemoglobin (< 9.0 gm/dL), or platelet count (100 K or >500 K) as evidenced by laboratory test results at Screening.
7. Any other active cause of optic neuropathy (Vitamin B12 deficiency, Vitamin E deficiency, etc.) or cardiac disease
8. EF less than 35% at last echocardiographic evaluation
9. Uncontrolled arrhythmia
10. Current use of any systemic chronic immunosuppressive drugs
11. Current use of Metformin

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Lynch, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia - Neurology, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 20 enrolled participants, 4 subjects screen failed and did not meet the study inclusion criteria. Of the 16 subjects who received treatment and 8 subjects withdrew after consenting and starting treatment from the study. 8 subjects completed all study visits.
Period: Overall Study
Arm/Group | Low Dose (20-30mg) | High Dose (40-60 mg)
Started | 8 | 8
Completed | 4 | 4
Not Completed | 4 | 4
Not completed — Lack of Efficacy | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Population: Of the 20 enrolled participants, 4 subjects screen failed and did not meet the study inclusion criteria. Of the 16 subjects who received treatment and 8 subjects withdrew after consenting and starting treatment from the study. 8 subjects completed all study visits.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose (20-30mg) | High Dose (40-60 mg) | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Customized [Count of Participants; unit: Participants]
  18-24 (years) | 3 | 2 | 5
  25-34 (years) | 2 | 2 | 4
  35-44 (years) | 2 | 2 | 4
  45-54 (years) | 0 | 2 | 2
  55-64 (years) | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 2 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 8 | 14
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in High Contrast Visual Acuity
Description: Change in High Contrast Visual Acuity will be measured by assessing the differences in the number of letters read (binocular) on the ETDRS High Contrast Visual Acuity Chart between groups (low dose and high dose).
Time Frame: Baseline to 52 weeks
Population: 2 subjects in low dose and 1 subject in the high dose did not complete Week 52 study visit
Measure: Median (Inter-Quartile Range); unit: Number of Letters Read on a Vision Board
Arm/Group | Low Dose (20-30mg) | High Dose (40-60 mg)
Number analyzed (Participants) | 6 | 7
Number of Letters Read on a Vision Board | 5.5 [0 to 6] | 0 [-5 to 6]

2. Secondary Outcome: Change in Low Contrast Visual Acuity
Description: Change in Low Contrast Visual Acuity will be measured by assessing the differences in the number of letters read (binocular) on the ETDRS Low Contrast Visual Acuity Chart between groups (low dose and high dose).
Time Frame: Baseline to 52 weeks
Population: All subjects in both low dose and high dose were unable to read a single letter on the low contrast vision board
Measure: Median (Inter-Quartile Range); unit: Number of Letters Read on a Vision Board
Arm/Group | Low Dose (20-30mg) | High Dose (40-60 mg)
Number analyzed (Participants) | 6 | 7
Number of Letters Read on a Vision Board | 0 [0 to 0] | 0 [0 to 0]

3. Secondary Outcome: Change in Low Luminescence Visual Activity
Description: Change in Low Luminescence Visual Acuity will be measured by assessing the difference in the number of letters read (binocular) on the ETDRS High Contrast Visual Acuity Chart with Low Luminescence Filter between groups (low dose and high dose).
Time Frame: Baseline to 52 weeks
Population: 2 subjects in low dose and 1 subject in the high dose did not complete Week 52 study visit
Measure: Median (Inter-Quartile Range); unit: Number of Letters Read on a Vision Board
Arm/Group | Low Dose (20-30mg) | High Dose (40-60 mg)
Number analyzed (Participants) | 6 | 7
Number of Letters Read on a Vision Board | 0.5 [0 to 2] | 0 [0 to 0]

4. Secondary Outcome: Change in Retinal Nerve Fiber Layer by Optical Coherence Tomography (OCT)
Description: The change in thickness of the retinal nerve fiber layer between groups (low dose and high dose) will be measured using the OCT, a non-invasive imaging test that uses light waves to take cross-section pictures of the retina.
Time Frame: Baseline to 52 weeks
Population: 6 low-dose and 7 high-dose subjects attempted to complete this procedure. However, due to disease progression (abnormal eye movements) and visual impairment (unable to focus on visual target) subjects were unable to perform the OCT exam in both low dose and high dose, thus resulting in poor quality images that were unable to be analyzed and will never be analyzed in the future.
Measure: Median (Inter-Quartile Range); unit: micron
Arm/Group | Low Dose (20-30mg) | High Dose (40-60 mg)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Visual Quality of Life by Visual Functioning Questionnaire (VFQ)
Description: The VFQ is a 25-item patient reported outcome on visual symptomology to assess change in patient self-report of visual ability over time compared to baseline between groups (low dose and high dose). The VFQ-25 consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. Each item is then converted to a 0 to 100 scale. The summary statistic is the difference in mean values from Baseline to Week 52. A negative value represents a worsening over time and a positive value represents improvement.
Time Frame: Baseline to 52 weeks
Population: 2 subjects in low dose and 1 subject in the high dose did not complete Week 52 study visit
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Low Dose (20-30mg) | High Dose (40-60 mg)
Number analyzed (Participants) | 6 | 7
Units on a scale | -2.42 (3.85) | 2.08 (5.77)

6. Secondary Outcome: Change in Cardiac Strain
Description: The change in cardiac strain (dL/L) in each dimension per cardiac cycle between groups (low dose and high dose) is measured by speckle tracking on imaging.
Time Frame: Baseline to 36 weeks
Population: Due to insufficient number of high quality reproducible scans we were unable to conduct a systematic analysis. The speckle tracking needed for this analysis was not done because reproducible scans were unobtainable in individuals with advanced FA due to inability to lie still for sufficient amounts of time and will never be analyzed in the future.
Measure: Mean (Standard Deviation)
Arm/Group | Low Dose (20-30mg) | High Dose (40-60 mg)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Cardiac Fibrosis
Description: The change in cardiac fibrosis over time by T1 mapping using late gadolinium enhancement between groups (low dose and high dose).
Time Frame: Baseline to 36 weeks
Population: Due to insufficient number of high quality reproducible scans we were unable to conduct a systematic analysis. The T1 mapping using late gadolinium enhancement needed for this analysis was not done because reproducible scans were unobtainable in individuals with advanced FA due to inability to lie still for sufficient amounts of time and will never be analyzed in the future.
Arm/Group | Low Dose (20-30mg) | High Dose (40-60 mg)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change Cardiac Stroke Volume
Description: The change in stroke volume will be calculated by Ejection Fraction x Ventricular Volume x Pulse Rate, over time between groups (low dose and high dose).
Time Frame: Baseline to 36 weeks
Population: 2 subjects in low dose and 2 subject in the high dose did not complete cardiac testing at the Week 36 study visit
Measure: Mean (Standard Deviation); unit: percentage of change in stroke volume
Arm/Group | Low Dose (20-30mg) | High Dose (40-60 mg)
Number analyzed (Participants) | 6 | 6
percentage of change in stroke volume | 0.12 (0.16) | -0.02 (0.29)

ADVERSE EVENTS:
Time Frame: AE's were assessed for approximately 104 weeks (2 years).
Description: The same subject reported both the pneumonia and pulmonary embolism SAEs.
Arm/Group | Low Dose (20-30mg) | High Dose (40-60 mg)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/8 | 2/8
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (20-30mg) (N=8) | High Dose (40-60 mg) (N=8)
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute Perforated Appendicitis (Surgical and medical procedures) | 0 (0) | 1 (3)
Vasovagal Episode (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (20-30mg) (N=8) | High Dose (40-60 mg) (N=8)
Injection Site Reaction: Pain, Tenderness, or Burning (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Injection Site Reaction: Erythema or Redness (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (6)
Injection Site Reaction: Induration or Swelling (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6)
Injection Site Reaction: Pruritus or Itching (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (6)
Injection Site Reaction: Urticaria or Hives (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Injection Site Reaction: Bruising (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Injection Site Reaction: Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Increased Bowel Frequency (Gastrointestinal disorders) | 1 (1) | 0 (0)
Viral Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Increased Appetite (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weight Gain (>10% of Body Weight) (Gastrointestinal disorders) | 1 (1) | 1 (1)
Weight Loss (<10% of Body Weight) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Edema (Vascular disorders) | 3 (3) | 0 (0)
Mucocele (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Increased Fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sore Throat (Infections and infestations) | 1 (1) | 0 (0)
Fever (Immune system disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 2 (2)
Viral Rhinitis or Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Altered Mental Status (Psychiatric disorders) | 2 (2) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 5 (5)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Black Eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chipped Teeth (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ear Infection (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Lactic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metallic Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Photosensitivity or Photodermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 1 (2) | 0 (0)
Blisters on Feet (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Leg Infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT05168774/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT05168774/ICF_001.pdf